CLINICAL TRIAL: NCT03664180
Title: Randomized Comparison of Anticoagulation After Primary Percutaneous Coronary Intervention Using Enoxaparin, ACT Guided Unfractionated Heparin or Bivalirudin Prolongation vs. no Anticoagulation To Improve Clinical Outcome
Brief Title: Comparison of Anticoagulation Prolongation vs. no Anticoagulation in STEMI Patients After Primary PCI
Acronym: RIGHT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Beijing Anzhen Hospital (Other)
Collaborators: Chinese Academy of Medical Sciences, Fuwai Hospital (Other); ACTION Study Group (Pitié-Salpêtrière Hospital), Paris, France (Unknown)
Responsible Party: Principal Investigator, Shao-Ping Nie, Professor of Medicine, Director, Emergency & Critical Care Center, Beijing Anzhen Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2018024X; BJUHFRIGHT201802 (Other: Beijing United Heart Foundation)
Record Dates: First submitted 2018-08-27; First posted 2018-09-10 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: STEMI - ST Elevation Myocardial Infarction
Keywords: anticoagulantion; post-procedure; STEMI
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — bivalirudin; Enoxaparin; Heparin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- anticoagulation (Experimental)
  Interventions: Drug: Bivalirudin; Drug: Enoxaparin; Drug: Unfractionated heparin
- No anticoagulation (Placebo Comparator)
  Interventions: Drug: Bivalirudin placebo; Drug: Enoxaparin placebo syringe; Drug: Unfractionated heparin placebo

INTERVENTIONS:
Drug: Bivalirudin — IV infusion of 0.2 mg/kg/h (low-rate infusion) for at least 48h after the procedure or until discharge from CCU if it occurs later
  Arms: anticoagulation
Drug: Enoxaparin — 40mg/d s.c.for at least 48h after the procedure or until discharge from CCU if it occurs later
  Arms: anticoagulation
Drug: Unfractionated heparin — IV infusion of 10 U/kg/h (maximum 1000 U) initially, adjusted to maintain ACT between 150 and 220 seconds for at least 48h after the procedure or until discharge from CCU if it occurs later
  Arms: anticoagulation
Drug: Bivalirudin placebo — Matching placebo IV infusion for at least 48h after the procedure or until discharge from CCU if it occurs later
  Arms: No anticoagulation
Drug: Enoxaparin placebo syringe — Placebo syringe will be only prepared by a designated unblended medical professional on site. Placebo syringe will be presented in identical containers as a clear, colorless, sterile liquid of saline.Subcutaneous injection once a day for at least 48 hours after the procedure or until discharge from CCU if it occurs later.
  Arms: No anticoagulation
Drug: Unfractionated heparin placebo — Matching placebo IV infusion for at least 48h after the procedure or until discharge from CCU if it occurs later.
  Arms: No anticoagulation

SUMMARY:
The RIGHT study is a large randomized study dedicated to post-PPCI anticoagulation in STEMI patients. The investigators propose to evaluate the clinical efficacy and safety of anticoagulation prolonged for at least 48 hours after the procedure vs. no prolongation of anticoagulation after procedure in patients with STEMI treated with bivalirudin during PPCI (primary hypothesis). When allocated to anticoagulation prolongation by randomization, the subject will be assigned to UFH, enoxaparin or bivalirudin (same regimen allocated by centre) for at least 48 hours after PPCI. The results from this study are expected to provide guidance on the risk/benefit of post-procedural anticoagulation in patients with STEMI.

DETAILED DESCRIPTION:
A minor change of time of randomization after prolongation of bivalirudin infusion at PCI dose up to 4 hours on protocol at September 19,2018. Reasons: a minor change concerning the timing of randomization considering the current local practice in some centers that use the 4 hour infusion of bivalirudin just after PCI. It remains in agreement with the current international guidelines and with the drug label in China. There is no change in drugs used and doses of these drugs once the randomization occurs.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old
* STEMI with PPCI of culprit lesion
* Bivalirudin therapy during PPCI
* Signed informed consent form

Exclusion Criteria:

* Patients with a formal indication for anticoagulation after PPCI (e.g. atrial fibrillation, left-ventricular thrombus, intra-aortic balloon pump, pulmonary embolism, mechanical heart valve)
* Patients with any indication for chronic anticoagulation
* Patient with previous lytic treatment
* Patient with previous coronary artery bypass graft surgery
* Cardiogenic shock, malignant ventricular arrhythmia, or mechanical complications
* Any anticoagulation other than bivalirudin started after the procedure before randomization
* Estimated body weight of >120 kg or <45kg
* BP ≥180/110mmHg at randomization
* Any bleeding diathesis or severe hematologic disease or history of intracerebral mass, aneurysm, arteriovenous malformation, recent (<6months) ischemic stroke or TIA, recent (<6months) intracranial hemorrhage or, gastrointestinal or genitourinary bleeding within the past 2 weeks
* History of heparin-induced thrombocytopenia
* Suspected acute aortic dissection (AAD)
* Major surgery within 1 month
* A planned elective surgical procedure that would necessitate an interruption in treatment with P2Y12 inhibitors in the next 6 months after enrollment
* Known PLT≤100×109 or HGB≤10g/L
* Known transaminase >3-fold ULN, or CCr<30ml/min
* Known allergy to any study drug
* Pregnancy or lactation
* Noncardiac coexisting conditions that could limit life expectancy to less than 1 year
* Current participation in an investigational drug or device trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2989 (Actual)
Dates: Start 2019-01-11 (Actual); Primary Completion 2022-11-23 (Actual); Study Completion 2022-11-23 (Actual)

PRIMARY OUTCOMES:
Primary efficacy endpoint - number of event of a composite of all-cause death, non-fatal myocardial infarction, non-fatal stroke, stent thrombosis (definite) or urgent revascularization (any vessel) | 30 days
  The number of event of a composite of all-cause death, non-fatal myocardial infarction, non-fatal stroke, stent thrombosis (definite) or urgent revascularization (any vessel) within 30 days after randomization
Primary safety endpoint - The number of event of major bleeding | 30 days
  The number of event of major bleeding (BARC 3 to 5) within 30 days after randomization

SECONDARY OUTCOMES:
Secondary ischemic endpoints - The number of event of a composite of all-cause death, non-fatal myocardial infarction, or non-fatal stroke | 30 days
  The number of event of a composite of all-cause death, non-fatal myocardial infarction, or non-fatal stroke within 30 days after randomization
Secondary ischemic endpoints - The number of event of a composite of all-cause death or non-fatal myocardial infarction | 30 days
  The number of event of a composite of all-cause death or non-fatal myocardial infarction within 30 days after randomization
Secondary ischemic endpoints - The number of cardiovascular death events | 30 days
  The number of cardiovascular death event within 30 days after randomization
Secondary ischemic endpoints - The number of stent thrombosis (ARC definite) events | 30 days
  The number of stent thrombosis (ARC definite) event within 30 days after randomization
Secondary safety endpoints - The number of bleeding events (TIMI, STEEPLE and GUSTO definition) | 30 days
  The number of bleeding events (TIMI, STEEPLE and GUSTO definition) within 30 days after randomization
  To demonstrate that post-procedure anticoagulation with UFH, enoxaparin or bivalirudin as compared to their placebo is associated to lower rate of the composite endpoint of major bleeding according to TIMI, STEEPLE and GUSTO definitions within the first 30 days after randomization.
Secondary safety endpoints - The number of thrombocytopenia events | 30 days
  The number of thrombocytopenia events within 30 days after randomization
  To demonstrate superiority of a strategy of post-procedure anticoagulation with UFH, enoxaparin or bivalirudin as compared to their placebo by the time from randomization to the first occurrence of any event of the Thrombocytopenia endpoint over 30 days of follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Anzhen Hospital, Capital Medical University, Beijing, China

REFERENCES:
- [Background] Yan Y, Wang X, Guo J, Li Y, Ai H, Gong W, Que B, Zhen L, Lu J, Ma C, Montalescot G, Nie S. Rationale and design of the RIGHT trial: A multicenter, randomized, double-blind, placebo-controlled trial of anticoagulation prolongation versus no anticoagulation after primary percutaneous coronary intervention for ST-segment elevation myocardial infarction. Am Heart J. 2020 Sep;227:19-30. doi: 10.1016/j.ahj.2020.06.005. Epub 2020 Jun 20. PMID 32663660
- [Derived] Yan Y, Guo J, Wang X, Wang G, Fan Z, Yin D, Wang Z, Zhang F, Tian C, Gong W, Liu J, Lu J, Li Y, Ma C, Vicaut E, Montalescot G, Nie S; RIGHT Investigators. Postprocedural Anticoagulation After Primary Percutaneous Coronary Intervention for ST-Segment-Elevation Myocardial Infarction: A Multicenter, Randomized, Double-Blind Trial. Circulation. 2024 Apr 16;149(16):1258-1267. doi: 10.1161/CIRCULATIONAHA.123.067079. Epub 2024 Feb 26. PMID 38406848